CLINICAL TRIAL: NCT05996692
Title: Evaluation of Adherence of Women With Fibromyalgia to Walking Prescriptions: a Cross-sectional Study
Brief Title: Evaluation of Adherence of Women With Fibromyalgia to Walking Prescriptions
Status: Completed | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Associate professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 39
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Walking; Adherence
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who walked regularly for exercise: Walking for exercise was explored according to a specific criterion (walking at least 30 min, in bouts of 15 min, with a small rest between bouts, twice a week, over a minimum of six consecutive weeks) based on previous recommendations.
  According to this criterion, the patients were divided into 2 groups as those who walked regularly for exercise and those who did not walk regularly for exercise.
  Interventions: Other: Evaluation of adherence to walking prescriptions
- Patients who did not walk regularly for exercise: Walking for exercise was explored according to a specific criterion (walking at least 30 min, in bouts of 15 min, with a small rest between bouts, twice a week, over a minimum of six consecutive weeks) based on previous recommendations.
  According to this criterion, the patients were divided into 2 groups as those who walked regularly for exercise and those who did not walk regularly for exercise.
  Interventions: Other: Evaluation of adherence to walking prescriptions

INTERVENTIONS:
Other: Evaluation of adherence to walking prescriptions — Adherence to walking prescriptions was evaluated according to a specific criterion (walking at least 30 min, in bouts of 15 min, with a small rest between bouts, twice a week, over a minimum of six consecutive weeks) based on previous recommendations.

SUMMARY:
Although there are many studies evaluating adherence to supervised walking programs in patients with fibromyalgia (FM), there are limited studies evaluating adherence to unsupervised walking programs.

DETAILED DESCRIPTION:
Although there are many studies evaluating adherence to supervised walking programs in patients with fibromyalgia (FM), there are limited studies evaluating adherence to unsupervised walking programs.

Purposes of this study were (1) to assess whether walking as exercise was prescribed by their physiatrist in Turkish women with FM who received pharmacological therapy, (2) to illustrate the frequency of patients who walk regularly as exercise, (3) to clinically compare patients who walk regularly as exercise and those who do not, and (4) to determine factors related to adherence to walking prescriptions.

ELIGIBILITY:
Inclusion Criteria:

* be between 18-70 years old
* female gender
* Pharmacological therapy has been recommended in the last 1 year

Exclusion Criteria:

* neurological disease or orthopedic problem presence that may be the reason of functional impairment
* neurological deficit presence

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since most of the patients with fibromyalgia are women, only female patients were included in the study, since a more homogeneous population was targeted.
Study Population: Patients diagnosed with FM according to the criteria of the American College of Rheumatology (ACR) and recommended pharmacological therapy within the last 1 year
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | through study completion, an average of one month
  Fibromyalgia Impact Questionnaire is a survey developed to measure functional status in FM patients. This scale measures 10 separate aspects, namely physical impairment, feel good, work missed, do job, pain, fatigue, rested, stiffness, anxiety, and depression. The total score in the questionnaire is between 0 and 100. Higher scores demonstrate higher disease severity and lower functional status.
The Tampa Scale for Kinesiophobia | through study completion, an average of one month
  The Tampa Scale for Kinesiophobia is a reliable survey on fear of movement. In the survey consisting of 17 questions, the total score is between 17 and 68, with higher scores indicating higher kinesiophobia.
Visual Analogue Scale | through study completion, an average of one month
  Overall pain intensity over the last 7 days was assessed with a Visual Analogue Scale (0 = no pain and 10 = the worst pain you can imagine).
Pain Catastrophizing Scale | through study completion, an average of one month
  Pain Catastrophizing Scale is made up of 13 items scored on a 5-point Likert scale from 0 (never) to 4 (always). The total score is obtained with the sum of the answers, being able to obtain a maximum score of 52. Higher scores in the scale represent a higher tendency to catastrophize.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Gaziler Physical Medicine and Rehabilitation Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No